CLINICAL TRIAL: NCT06421597
Title: Identifying Individuals At Risk of Glucocorticoid-Induced Impairment of Bone Disease
Acronym: RIGID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other); University of Ulm (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-506949-27-00
Record Dates: First submitted 2024-05-03; First posted 2024-05-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis Secondary
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone group (Experimental)
  Interventions: Drug: Prednisolone
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — prednisoline 25 mg/day for seven days
  Arms: Prednisolone group
Drug: Placebo — Placebo treatment for seven days
  Arms: Placebo group

SUMMARY:
Previous studies have shown that there is a large inter-individual variability in the degree of bone loss during glucocorticoid treatment, and while some patients experience extensive bone loss other patients' bone mass remains stable. The aim of the study is to find a biomarker that can be used to identify individuals at risk of glucocorticoid-induced bone loss. The study will include 36 healthy volunteers, that will be randomized to receive either glucocorticoid treatment or placebo. During the study blood samples, bone marrow samples, bone tissue samples, and adipose tissue samples are taken and an oral glucose tolerance test is performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-50 years.

Exclusion Criteria:

* Uncontrolled thyrotoxicosis
* Chronic kidney disease (eGFR <30)
* Known Cushing's syndrome
* Previous gastric bypass and/or known ongoing malabsorption
* Severe covid-19 in the last 3 month (defined as needing dexamethasone treatment)
* Use of oral or inhaled glucocorticoids within the past year
* Menopause (defined as 1 year without menstrual bleeding)
* Pregnancy (defined as elevated HCG)
* Ongoing infection
* Allergy to prednisolone or one of the excipients
* Systematic fungal infections
* Vaccination with living or weaken viral or bacterial vaccines in patient who or immunocompromised. In these cases, prednisolone treatment should not be administered two weeks before and after vaccination
* Not able to provide informed consent (e.g., dementia, not able to understand Danish).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Procollagen type 1 N-terminal propeptide (P1NP) | Baseline to day 8
  Changes in the level of the bone turnover marker P1NP in peripheral blood from baseline to day 8

SECONDARY OUTCOMES:
Collagen 1 cross link C-terminal telopeptide (CTX) | Baseline to day 8 and 15
  Changes in the level of the bone turnover marker CTX in peripheral blood from baseline to day 8 and 15
P1NP (baseline to day 15) | Baseline to day 15
  Changes in the level of the bone turnover marker P1NP in peripheral blood from baseline to day 15
Concentration of Glucocorticoid metabolites | Baseline to day 8
  Changes in the levels of glucocorticoid metabolites in blood from baseline to day 8
Adipose tissue | Baseline to day 8
  Changes in gene expression in abdominal and gluteal subcutaneous adipose tissue from baseline to day 8
Bone tissue | Baseline to day 8
  Changes in gene expression in bone tissue from baseline to day 8
Glucose | Baseline to day 8
  Changes in glucose levels during a mixed meal test from baseline to day 8
C-peptid | Baseline to day 8
  Changes in c-peptid levels during a mixed meal test from baseline to day 8

OTHER OUTCOMES:
Biomarker | Baseline
  Untargeted proteomics will be used to try to identify a biomarker for individuals at risk of glucocorticoid induced bone loss

CONTACTS AND LOCATIONS:
Overall Officials: Anja Lisbeth Frederiksen, MD, Principal Investigator — Odense University Hospital; Claus Bogh Juhl, MD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (2):
- Denmark (2):
  - Hospital of South West Jutland, Esbjerg
  - Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers other than collaborators. Since the data contains personal information from the study participants